CLINICAL TRIAL: NCT05784870
Title: A Multicenter Randomized Controlled Study of Shengxuening Tablet in the Treatment of Chemotherapy-related Anemia in Hematologic Tumors
Brief Title: A Study of Shengxuening Tablet in the Treatment of Chemotherapy-related Anemia in Hematologic Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Fuling Zhou, Head,Division of Hematology; Professor of Hematology; Doctoral advisor, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06
Record Dates: First submitted 2023-02-25; First posted 2023-03-27 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hematological Malignancy; Cancer-Related Anemia
Keywords: Shengxuening tablet; chemotherapy-related Anemia
MeSH Terms: conditions — Hematologic Neoplasms | interventions — shengxuening; ferrous succinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shengxuening Tablets (Experimental): Oral treatment with Shengxuening Tablets 1 week before chemotherapy, usage: 0.5gtid, for 28 consecutive days
  Interventions: Drug: Shengxuening Tablet
- ferrous succinate (Active Comparator): Oral treatment with ferrous succinate 1 week before chemotherapy, usage: 200mgqd, for 28 consecutive days
  Interventions: Drug: Ferrous succinate

INTERVENTIONS:
Drug: Shengxuening Tablet — Oral treatment with Shengxuening Tablets 1 week before chemotherapy, usage: 0.5gtid, for 28 consecutive days
  Arms: Shengxuening Tablets
Drug: Ferrous succinate — Oral treatment with ferrous succinate 1 week before chemotherapy, usage: 200mgqd, for 28 consecutive days
  Arms: ferrous succinate

SUMMARY:
Cancer-related anemia (CRA) is one of the common accompanying diseases of malignant tumors. In 2019, a cross-sectional survey on the anemia status of 7324 malignant tumor patients in 97 hospitals in China found that the incidence of CRA was about 49.24%. 92.84% of the patients have not been given enough attention and effective treatment. According to the European Oncological Anemia Survey, CRA has the highest incidence in leukemia patients, followed by lymphoma/myeloma. CRA not only leads to a decline in the quality of life of patients, but also reduces the sensitivity to radiotherapy and chemotherapy, and also causes hypoxia in tumor tissue, which affects the prognosis of patients as an independent factor. At present, the treatment of CRA mainly includes blood transfusion therapy, erythropoiesis-stimulating agent (ESA) therapy, iron supplementation, etc. Conventional oral iron has low bioavailability and strong gastrointestinal irritation. Although intravenous iron can quickly replenish iron, excessive iron supplementation is prone to iron overload. Less acceptable. Shengxuening Tablets are derived from silkworm excrement. The main components of iron chlorophyllin and chlorophyll derivatives are very similar in structure to heme, and can be directly absorbed by small intestinal mucosal cells, effectively supplementing the iron elements required in the process of hematopoiesis. The investigators found that Shengxuening Tablets can increase the number of peripheral blood cells in mouse models of myelosuppression, improve bone marrow morphology, reverse the decrease in body weight and spleen index, and increase the levels of serum erythropoietin and granulocyte-macrophage colony-stimulating factor . Real-time fluorescent quantitative PCR and Western blot analysis showed increased expression levels of stem cell factor (SCF), JAK2 and STAT3 in the liver. These results indicated that Shengxuening Tablets promoted the recovery of hematopoietic function in myelosuppressive models by increasing the secretion of hematopoietic factors and activating the JAK2/STAT3 pathway. Therefore, in order to further confirm the preventive effect, effectiveness and safety of Shengxuening Tablets in the treatment of anemia in patients with hematological tumors complicated with anemia, this clinical trial was designed.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old, gender is not limited;
* Patients diagnosed with blood cancer complicated with anemia;
* During the screening period of ≤1 week, hemoglobin (Hb): 60g/L<Hb≤100g/L;
* Willingness to treat

Exclusion Criteria:

* During the screening period of ≤1 week, hemoglobin (Hb)≤60g/L
* History of blood transfusion within 1 month;
* Urgent blood transfusion or EPO infusion is required within the screening period of ≤1 week;
* Folic acid or vitamin B12 deficiency;
* History of iron allergy, history of allergy or intolerance to the study drug;
* Pregnant and lactating women;
* Age <18 years old and body weight ≤35kg;
* Participated in other clinical drug research in the past 3 months;
* Severe cardiac insufficiency (NYHA grade III or above);
* Severe abnormal liver function (ALT, AST and TBIL ≥ 2 times the upper limit of normal value);
* Severe renal insufficiency (creatinine clearance ≤ 15ml/min);
* Severe mental disorder;
* Acute and chronic blood loss;
* Combined with a second tumor;
* Ferritin>500μg/L;
* Combined with active tuberculosis;
* Failure to cooperate with treatment according to doctor's advice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  Hemoglobin in g/L
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  Red Blood Cell in 10^12/L
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  mean corpuscular hemoglobin in pg
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  mean corpuscular volume in fL
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  Red blood cell specific volume in percentage
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  Reticulocyte in 10^9/L
Change from Blood routine in plasma at Week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  Serum erythropoietin in ng/ml

SECONDARY OUTCOMES:
Changes from iron metabolism indicators in plasma at week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  serum ferritin in μg/L
Changes from iron metabolism indicators in plasma at week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  serum iron in μmol/L
Changes from iron metabolism indicators in plasma at week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  total iron binding capacity in μmol/L
Changes from iron metabolism indicators in plasma at week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  unsaturated iron binding capacity in μmol/L
Changes from iron metabolism indicators in plasma at week 4 | Day 0，Week 1，Week2，Week 3，Week 4
  transferrin saturation in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided